CLINICAL TRIAL: NCT06942533
Title: The Effect of Visual Feedback From the SpiroGym Mobile Application on Expiratory Muscle Strength Training Performance in Patients With Parkinson's Disease
Brief Title: Effect of Visual Feedback From the SpiroGym Mobile Application
Acronym: EXPARK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Martin Srp, Ph.D., Chief physiotherapist, General University Hospital, Prague
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EXPARK
Record Dates: First submitted 2025-04-09; First posted 2025-04-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease; Breathing Exercises; Telemedicine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Each PD patient will complete two EMST sessions separated by a two-week period. One session will include feedback via the SpiroGym mobile application, while the other will be performed without such feedback. The order of these conditions will be randomly assigned. Patients cannot be fully blinded in this trial, as they may subjectively perceive differences between conditions. However, they will be partially blinded by withholding information about the study hypothesis. Patients will be informed only that the study compares different strategies for expiratory muscle training. If a patient asks which intervention is more effective, the examiner will respond that both methods are expected to be equally effective.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMST with video feedback via the SpiroGym mobile application (Experimental): Patients will complete one EMST session with the SpiroGym app.
  Interventions: Device: EMST with SpiroGym app
- EMST without video feedback via the SpiroGym mobile application (Active Comparator): Patients will complete one EMST session without the SpiroGym app.
  Interventions: Device: EMST without SpiroGym app

INTERVENTIONS:
Device: EMST with SpiroGym app — Participants will perform expiratory muscle training using an Expiratory Muscle Trainer (EMST150; Aspire Products, LLC, United States). Participants will be instructed to perform five sets of five forceful expirations coupled with the SpiroGym app.
  Video feedback via the SpiroGym app: During correct performance of the expiratory manoeuvre with the handheld device, the exhalation valve opens and the resulting airflow increases the sound level detected by the microphone. Simultaneously, the application provides real-time visual feedback on the mobile phone screen as a curve depicting the current sound level. The patient's task is to keep the curve within the training zone, defined by two lines corresponding to the lower and upper thresholds.
  Arms: EMST with video feedback via the SpiroGym mobile application
Device: EMST without SpiroGym app — Participants will perform expiratory muscle training using an Expiratory Muscle Trainer (EMST150; Aspire Products, LLC, United States). Participants will be instructed to perform five sets of five forceful expirations without the SpiroGym app.
  Arms: EMST without video feedback via the SpiroGym mobile application

SUMMARY:
The previous pilot study showed that two weeks of intensive expiratory muscle strength training (EMST) with SpiroGym was sufficient to significantly improve voluntary peak cough flow (PCF). The improvement was quantitatively comparable to that reported in other intensive EMST studies of longer duration. To explain this rapid improvement, we considered the potential contribution of SpiroGym's visual feedback. We assumed that real-time visual feedback increased training effort compared with conventional EMST performed without immediate feedback.

The aim of this study is to evaluate the effect of visual feedback provided by the SpiroGym mobile application on performance during expiratory muscle strength training in patients with Parkinson's disease.

DETAILED DESCRIPTION:
The study will be conducted using a prospective crossover design. Patients with Parkinson's disease will complete two EMST sessions, each at 75% of maximum expiratory pressure (MEP), separated by a two-week interval. One EMST session will include feedback via the SpiroGym mobile application, while the other will be performed without feedback. The order of these conditions will be randomly assigned.

Primary hypothesis

1. Visual feedback provided by the SpiroGym application during expiratory training will result in greater muscle activation, as measured by surface electromyography (sEMG), compared with training without visual feedback.

   Secondary hypotheses
2. Visual feedback during expiratory training will lead to greater expiratory performance, reflected by higher noise intensity recorded by the SpiroGym application, than training without visual feedback.
3. Participants will report lower perceived difficulty and higher motivation to perform expiratory training exercises when visual feedback is provided than when it is absent.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinsons disease
* Stable dopaminergic medication (stable dose for at least 1 month)

Exclusion Criteria:

* Other neurological disorders
* Significant cognitive impairment
* Major psychiatric disorder
* History of head or neck cancer or previous surgical interventions in the neck region.
* Illness during the study period

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Surphace elektromyography (sEMG) measurement of abdominal muscle (m. obliquus internus abdominis). | Baseline, week 2
  Wireless sEMG electrodes will be placed on the clean skin of the abdominal muscle (m. obliquus internus abdominis). A reference voluntary contraction (RVC) will be used to normalize the sEMG data. sEMG of the abdominal muscle (m. obliquus internus abdominis) during two conditions (EMST with SpiroGym and EMST without SpiroGym) will be compared.

SECONDARY OUTCOMES:
SpiroGym Sound Intenzity (SSI) measurement | Baseline, week 2
  The output from the SpiroGym application (SpiroGym Sound Intensity - SSI), which records the intensity of the sound generated by the expiratory device (note: the louder the sound, the greater the expiratory force) during two conditions (EMST with SpiroGym and EMST without SpiroGym) will be compared.
Surphace elektromyography (sEMG) measurement of suprahyoid muscle complex and abdominal muscles (m. rectus abdominis and m. obliquus externus abdominis). | Baseline, week 2
  Wireless sEMG electrodes will be placed on the clean skin of the suprahyoid muscle complex and abdominal muscle (m. rectus abdominis and m. obliquus externus abdominis). A reference voluntary contraction (RVC) will be used to normalize the sEMG data. sEMG of the suprahyoid muscle complex and abdominal muscle (m. rectus abdominis and m. obliquus externus abdominis) during two conditions (EMST with SpiroGym and EMST without SpiroGym) will be compared.
Participant's Feedback questionnaire | week 2
  After all the maneuvers were completed over the two sessions, participants will complete a questionnaire focused on the subjective perception of exercise difficulty and motivation to perform it with or without visual feedback. The questionnaire will be rated using a Likert scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - General University Hospital, Prague
  - Department of Neurology and Centre of Clinical Neuroscience First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Srp M, Bartosova T, Klempir J, Lagnerova R, Gal O, Listvanova T, Jech R, Ruzicka E, Hoskovcova M. Expiratory Muscle Strength Training in Multiple System Atrophy: A Pilot Study. Mov Disord Clin Pract. 2023 May 19;10(7):1060-1065. doi: 10.1002/mdc3.13765. eCollection 2023 Jul. PMID 37476315